CLINICAL TRIAL: NCT02810002
Title: Assessing Foot Injuries in Infantry Recruits Wearing Different Boots, a Prospective Randomized Study
Brief Title: Assessing Foot Injuries in Infantry Recruits Wearing Different Boots
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDF-1346-2014
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Blister; Abrasion; Stress Fracture; Ankle Sprain; Patellofemoral Pain Syndrome; Back Pain
MeSH Terms: conditions — Blister; Fractures, Stress; Ankle Injuries; Patellofemoral Pain Syndrome; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DEFINITE-REGULATOR (Experimental): Training with DEFINITE-REGULATOR experiment infantry boots manufactured by Brill Industries, Rishon LeZion, Israel
  Interventions: Device: Experimental infantry boot - DEFINITE-REGULATOR
- modified Belleville 390 TROP (Active Comparator): Standard issue infantry boot
  Interventions: Device: Control infantry boot

INTERVENTIONS:
Device: Experimental infantry boot - DEFINITE-REGULATOR — Training: infantry basic training in the experimental boots
  Arms: DEFINITE-REGULATOR
Device: Control infantry boot — Training: infantry basic training in the control boots
  Arms: modified Belleville 390 TROP

SUMMARY:
One hundred infantry recruits will be randomly assigned to two groups. Injuries will be monitored.

DETAILED DESCRIPTION:
One hundred infantry recruits will be randomly assigned to receive experimental infantry boots (DEFINITE-REGULATOR) or standard issued boots (modified Belleville 390 TROP).

Overuse injuries and foot injuries will be monitored over a period of 14 weeks. The intervention group will wear experimental infantry boots and the controls will wear standard issue boots.

ELIGIBILITY:
Inclusion Criteria:

* Infantry recruits on selected base

Exclusion Criteria:

* None

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of recruits with at least one injury related to the boots | 14 weeks
  Injuries assessed: Blister, Abrasion, Stress Fracture, Ankle Sprain, Patellofemoral Pain Syndrome, Back Pain

IPD SHARING:
Plan to Share IPD: Yes
Raw unidentified data available by contacting the PI

REFERENCES:
- [Derived] Milgrom C, Sorkin A, Gam A, Singer J, Nir I, Kogan B, Finestone AS. The search for the best infantry boot. Disaster Mil Med. 2016 Oct 10;2:14. doi: 10.1186/s40696-016-0024-5. eCollection 2016. PMID 28265448